CLINICAL TRIAL: NCT05234606
Title: A Phase 1/2, Open-Label, Dose-Escalation and Expansion Study of SBT6290 Alone and in Combination With PD-(L)1 Inhibitors in Subjects With Advanced Solid Tumors Associated With Nectin-4 Expression
Brief Title: A Safety and Preliminary Efficacy Study of SBT6290 Alone and in Combination With PD-(L)1 Inhibitors in Select Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on strategic re-alignment
Sponsor: Silverback Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBT6290-101
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Urothelial Carcinoma; Triple Negative Breast Cancer; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Hormone Receptor-positive/HER2-negative Breast Cancer
Keywords: SBT6290; breast cancer; urothelial carcinoma; non-small cell lung cancer; squamous cell carcinoma of head and neck; TLR8; Nectin-4; pembrolizumab (KEYTRUDA)
MeSH Terms: conditions — Carcinoma, Transitional Cell; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: SBT6290 (Experimental): SBT6290 every 3 weeks
  Interventions: Drug: SBT6290
- Part 2: SBT6290 (Experimental): SBT6290 every 3 weeks
  Interventions: Drug: SBT6290
- Part 3: SBT6290 + pembrolizumab (Experimental): SBT6290 plus pembrolizumab every 3 weeks
  Interventions: Drug: SBT6290; Drug: pembrolizumab
- Part 4: SBT6290 + pembrolizumab (Experimental): SBT6290 plus pembrolizumab every 3 weeks
  Interventions: Drug: SBT6290; Drug: pembrolizumab

INTERVENTIONS:
Drug: SBT6290 — Escalating doses by subcutaneous (SC) injection in 21-day cycles
  Arms: Part 1: SBT6290; Part 3: SBT6290 + pembrolizumab
Drug: SBT6290 — Dose expansion with the recommended Phase 2 dose (RP2D) by SC injection in 21-day cycles
  Arms: Part 2: SBT6290; Part 4: SBT6290 + pembrolizumab
Drug: pembrolizumab — 200 mg via intravenous (IV) injection in 21-day cycles
  Other Names: KEYTRUDA
  Arms: Part 3: SBT6290 + pembrolizumab; Part 4: SBT6290 + pembrolizumab

SUMMARY:
This is a first-in-human, open-label, multicenter, dose-escalation and expansion study designed to investigate SBT6290 administered alone and in combination with pembrolizumab in advanced solid tumors associated with Nectin-4 expression.

DETAILED DESCRIPTION:
This is a first-in-human study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, immunogenicity, and preliminary antitumor activity of SBT6290 administered subcutaneously (SC) as a monotherapy and in combination with pembrolizumab in solid tumors associated with Nectin-4 expression. There are 4 parts to this study:

* Part 1: A dose escalation of SBT6290 monotherapy
* Part 2: Tumor-specific expansion cohorts evaluating SBT6290 monotherapy administered at the recommended phase 2 dose (RP2D) identified in Part 1
* Part 3: A dose escalation of SBT6290 in combination with pembrolizumab
* Part 4: An expansion cohort of SBT6290 in combination with pembrolizumab administered at the RP2D identified in Part 3 for the combination

ELIGIBILITY:
Key Inclusion Criteria:

* Locally advanced or metastatic solid tumors associated associated with Nectin-4 expression (locally advanced or metastatic urothelial carcinoma, TNBC, NSCLC, SCCHN, and HR+/HER2- negative breast cancer)
* Measurable disease per the the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria
* Tumor lesion amenable for biopsy available to submit for retrospective baseline testing of Nectin-4; archived tumor tissue may be acceptable depending upon study Part detailed criteria
* ECOG Performance Status of 0 or 1
* Adequate organ and marrow function Note: Other protocol-defined inclusion/exclusion criteria may apply.

Key Exclusion Criteria:

* History of allergic reactions to certain components of study treatments
* Untreated brain metastases
* Currently active (or history of) autoimmune disease
* Taking the equivalent of >10 mg / day of prednisone
* Uncontrolled or clinically significant interstitial lung disease (ILD)
* History of ongoing, uncontrolled, symptomatic eye disorders requiring intervention or associated with marked visual field defects or limiting age-appropriate instrumental activities of daily living
* HIV infection, active hepatitis B or hepatitis C infection Note: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities: Part 1 and Part 3 | Up to 28 days after the first dose of SBT6290
  Severity of treatment-emergent adverse events as assessed by the NCI CTCAE Version 5.0.
Number of Participants With Treatment-emergent Adverse Events: All Parts | From enrollment to 30 days after the last dose of SBT6290, up to 2 years
  Severity of treatment-emergent adverse events as assessed by the NCI CTCAE Version 5.0.
Number of Participants With an Objective Response Rate: Part 2 and Part 4 | From enrollment to confirmed response, up to 1 year
  Complete response and partial response as assessed by RECIST Version 1.1 Criteria.
Duration of Response for Participants With an Objective Response Rate: Part 2 and Part 4 | From enrollment until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 3 years
  Complete response and partial response as assessed by RECIST Version 1.1 Criteria.

SECONDARY OUTCOMES:
Number of Participants With an Objective Response Rate: Part 1 and Part 3 | From enrollment to confirmed response, up to 1 year
  Complete response and partial response as assessed by RECIST Version 1.1 Criteria.
Duration of Response for Participants With an Objective Response Rate: Part 1 and Part 3 | From enrollment until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 3 years
  The length of time from the participant's first complete response or partial response as assessed by RECIST Version 1.1 Criteria until disease progression or death.
Rate of Disease Control for Participants: All Parts | Up to at least 6 months after the first dose of SBT6290
  Complete response, partial response, and stable disease as assessed by RECIST Version 1.1 Criteria.
Progression-free Survival: Part 2 | From first dose of SBT6290 until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 3 years
  Complete response, partial response, stable disease, and progressive disease as assessed by RECIST Version 1.1 Criteria.
Estimates of Selected PK Parameters for SBT6290: All Parts | Immediately before and after SBT6290 doses up to 2 years
  Maximum concentration (Cmax).
Estimates of Selected PK Parameters for SBT6290: All Parts | Immediately before and after SBT6290 doses up to 2 years
  Area under the plasma concentration versus time curve (AUC).
Incidence of SBT6290 Antidrug Antibodies (ADA): All Parts | Immediately before and after SBT6290 doses for up to 2 years
  Number of participants positive for ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Angra, PharmD, Study Director — Silverback Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu F, Xu K, Fan L, Li X, Liu Y, Yang F, Zhu C, Guan X. Estrogen receptor beta suppresses the androgen receptor oncogenic effects in triple-negative breast cancer. Chin Med J (Engl). 2024 Feb 5;137(3):338-349. doi: 10.1097/CM9.0000000000002930. Epub 2023 Dec 15. PMID 38105538